CLINICAL TRIAL: NCT06953375
Title: Implementation of Neuromuscular Electrical Stimulation After Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Colorado Health (Other); Intermountain Health Care, Inc. (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-0868; R01AG084683 (NIH)
Record Dates: First submitted 2024-11-21; First posted 2025-05-01 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Total Knee Arthroplasty; Functional Recovery; Aging; Physical Therapy
Keywords: NMES (Neuromuscular Electrical Stimulation); TKA (Total Knee Arthroplasty); Rehabilitation; Physical Therapy; RE-AIM: Reach Effectiveness Adoption Implementation Maintenance; Implementation Science; Older Adults; Physical Function

STUDY DESIGN:
Who Masked: Participant
Masking Description: Investigators will not be blinded to the arms due to facility/clinician training required for this study design. Study sites (i.e., outpatient physical therapy clinics) will be the unit of randomization. Study sites will be made broadly aware of the study initiative during the site recruitment process; however, the site will not be provided with detailed information about the intervention unless randomized to the Intervention arm. As such, clinicians, or rehabilitation care providers, at usual care sites will remain blinded to the intervention for the duration of the study. Clinicians will collect patient-level functional outcomes as part of their standard of care and all patients who are subjects of the intervention will not be aware of the group allocation in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NMES (Experimental): Neuromuscular Electrical Stimulation (NMES) consists of usual care rehabilitation plus evidence-based implementation of NMES in the early postoperative period to improve physical function after TKA.
  Interventions: Procedure: NMES
- Usual Care (Active Comparator): The Usual Care clinics will continue clinical practice as normal. Usual Care sites will not have overlap of personnel or training with NMES Sites.
  Interventions: Other: Usual Care

INTERVENTIONS:
Procedure: NMES — The NMES intervention protocol in this study ensures patients receive NMES intervention that is adequately dosed (dose = treatment minutes x intensity), delivered using evidence-based parameters, and feasible. The investigators will deliver NMES using a portable two-channel stimulator that the investigators have found to produce stronger muscle contractions than other portable NMES units and has been used in previous clinical studies. It also has a built-in compliance meter to monitor patient treatment minutes (adherence) to NMES application. NMES sites will perform routine collection of outcomes as part of standard practice.
  Arms: NMES
Other: Usual Care — Usual Care clinics will continue with routine collection and documentation of physical performance outcomes as standard practice. A combination of chart reviews and on-site or remote observation will allow for characterization of usual care components for descriptive comparison. Usual Care clinics including the facility, rehabilitation clinicians, and patients will not have access to NMES materials developed for this study.
  Arms: Usual Care

SUMMARY:
Patients experience dramatic quadriceps strength loss after total knee replacement, which contributes to persistent weakness and reduced long-term function after surgery. Neuromuscular electrical stimulation (NMES) reduces quadriceps weakness and improves patient function after knee replacement, but it is drastically underused in rehabilitation practice. This randomized trial will examine the effectiveness and feasibility of a comprehensive strategy for implementing neuromuscular electrical stimulation after knee replacement in two large healthcare organizations.

DETAILED DESCRIPTION:
Total Knee Arthroplasty (TKA) reduces pain and disability caused by knee osteoarthritis, but the surgery results in substantial trauma to the knee. This acute trauma exacerbates underlying weakness-especially in the quadriceps. This leads to muscle atrophy and likely contributes to the long-term weakness and disability patients with TKA experience relative to their healthy peers. Attenuating quadriceps strength loss should be a primary target for improving rehabilitation outcomes after TKA.

Neuromuscular electrical stimulation (NMES) is recommended in TKA clinical practice guidelines to attenuate quadriceps strength loss. In controlled settings, NMES has established efficacy and attenuates quadriceps strength loss by 40% in the first month after surgery by overriding muscle activation deficits and reducing muscle atrophy. However, the effectiveness of NMES after TKA has not been adequately studied in real-world clinical settings, and preliminary data suggests that less than 4% of rehabilitation clinicians are using NMES as recommended by current TKA practice guidelines.

To address this gap, the investigators will conduct a cluster randomized trial in two healthcare systems (UCHealth and Intermountain Health) and their associated outpatient physical therapy clinics (n=30) to evaluate the effectiveness and implementation of NMES to address musculoskeletal deficits after TKA.

The investigators will compare outcomes between patients who receive contemporary rehabilitation supported by a comprehensive NMES implementation strategy (NMES) to patients who receive contemporary musculoskeletal rehabilitation alone (Usual Care; Aim 1). The investigators will gather information on NMES implementation to promote its uptake and translation to clinical practice (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

Site Inclusion Criteria:

• UCHealth or Intermountain Health outpatient physical therapy clinic

Patient Inclusion Criteria:

* Underwent primary unilateral TKA
* Attended outpatient rehabilitation at a participating clinic within 5 days after TKA
* Attended at least 3 total outpatient physical therapy visits in total

Exclusion Criteria:

Patient Exclusion Criteria:

* NMES Contraindications [Patients with implanted cardiovascular cardiovertedefibrillator (ICD), active cancer, post-operative diagnosed deep vein thrombosis (DVT) in involved lower extremity]
* Previous lower extremity arthroplasty less than 12 weeks prior to scheduled TKA surgical date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3250 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) | Pre-operative visit; Post-operative PT baseline, 2 weeks, 4 weeks (primary endpoint), 6 weeks, up to 24 weeks
  The TUG is a measure of mobility and balance that consists of rising from a seated position, walking three meters, and pivoting and returning to the original seated position. Faster times indicate better physical function.

SECONDARY OUTCOMES:
30 Second Sit-to-Stand (30-STS) | Pre-operative visit; Post-operative PT baseline, 2 weeks, 4 weeks (primary endpoint), 6 weeks, up to 24 weeks
  The 30-STS is a measure of lower body strength and stamina that consists of moving from sitting to a full stand as many times as possible in 30 seconds. More completions indicate better physical function.
Quadriceps Strength | Pre-operative visit; Post-operative PT baseline, 2 weeks, 4 weeks (primary endpoint), 6 weeks, up to 24 weeks
  A commercially available hand dynamometer that uses a Bluetooth-enabled tensile load sensor will be used to assess quadriceps strength. Load sensors are reliable and valid for assessing isometric quadriceps strength. Higher scores indicate more strength
Knee Outcome Survey Activities of Daily Living Scale (KOS-ADL) | Pre-operative visit; Post-operative PT baseline, 2 weeks, 4 weeks (primary endpoint), 6 weeks, up to 24 weeks
  The Knee Outcome Survey Activities of Daily Living Scale (KOS-ADL) provides a score of patients' self-reported knee stiffness, pain, and function. Scores range from 0% to 100%, with higher scores indicating fewer symptoms affecting activities of daily living.
Knee Range of Motion (ROM) | Pre-operative visit; Post-operative PT baseline, 2 weeks, 4 weeks (primary endpoint), 6 weeks, up to 24 weeks
  ROM measures the amount of movement a joint can make in a specific direction and will be assessed using a goniometer. Higher degrees of movement indicate better range of motion.
Visit Utilization | Post-operative PT baseline up to 24 weeks
  Visit utilization will be defined as the number of outpatient physical therapy visits attended during the patient's postoperative rehabilitation episode-of-care.
Patient Satisfaction | Post-operative 6 weeks
  A self-report satisfaction survey will be administered. Patient Satisfaction consists of items rated on a 5-point Likert scale. Higher scores indicate better satisfaction.
NMES Satisfaction | Post-operative 6 weeks
  NMES Satisfaction is a self-report survey and consists of items rated on a 5 point Likert scale. Higher scores indicate better satisfaction.

OTHER OUTCOMES:
NMES Intensity | Post-operative PT baseline, 2 weeks, 4 weeks (primary endpoint), 6 weeks, up to 24 weeks
  The magnitude of NMES-induced muscle contraction elicited by patient.
NMES Adherence | Post-operative week 6
  The proportion of prescribed NMES minutes completed by a patient will be measured by NMES unit.
RE-AIM Reach | Throughout experimental phase (about 2.5 years)
  Proportion of patients treated with NMES out of all eligible patients
RE-AIM Adoption | Throughout experimental phase (about 2.5 years)
  Proportion of clinicians using NMES with at least 80% of eligible patients out of all trained clinicians at intervention clinics.
RE-AIM Implementation | Throughout experimental phase (about 2.5 years)
  Proportion of prescribed NMES time (15 mins, twice per day) completed by patient (measured by NMES unit) over the course of the study.
RE-AIM Maintenance | 6 months following end of experimental phase
  Proportion of clinicians using NMES with at least 80% of eligible patients out of all trained clinicians at intervention clinics.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Stevens-Lapsley, PT, PhD, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - UCHealth, Aurora, Colorado
  - University of Colorado Denver, Anschutz, Aurora, Colorado
  - Intermountain Health, Murray, Utah

IPD SHARING:
Plan to Share IPD: Yes
The study team guarantees that all data collected as part of this project will be released in accordance with standard data sharing policies and procedures to validate research findings if requested. Data will be made available in a timely manner to the broader scientific community, and will be complete, and as accurate as possible. All data released will be de-identified, with no information that could be linked to any study subjects, or participating study practices to ensure the confidentiality of all subjects and practices. If necessary, a data use agreement will be established.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be made available 12 months after primary study publication
Access Criteria: Data will be made available upon reasonable written request to the study team. The PI, Dr. Jennifer Stevens-Lapsley will review requests.